CLINICAL TRIAL: NCT06876025
Title: Activities and Social Participation of Children With Atypical Motor Development
Brief Title: Children's Activities and Social Participation
Status: Completed | Type: Observational
Sponsor: Federal Institute of Rio de Janeiro (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Elisa Beatriz van Eyken, PhD Professor, Federal Institute of Rio de Janeiro
Other Study IDs: 559; CAAE 59793122.8.0000.5268 (Other: Research Ethics Committee)
Record Dates: First submitted 2023-06-06; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Child Development Disorder
Keywords: ICF; Child development; Social participation; Child
MeSH Terms: conditions — Developmental Disabilities | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Caregivers: Caregivers will respond to two of the three questionnaires: PEM-CY or YC-PEM, and PEDI
  Interventions: Other: questionnaires

INTERVENTIONS:
Other: questionnaires — Application of the questionnaires Measure of Participation and Environment - Children and Youth, (PEM-CY), or Measure of Participation and the environment - young children (YC-PEM), and the Pediatric Disability Assessment Inventory (PEDI).

SUMMARY:
The goal of this observational study is to learn the perception of caregivers about the limitations of activities, and the restriction in the social participation of children who are in Neurofunctional physiotherapy. The main questions it aims to answer are:

* What is the ability to perform tasks, and
* how is the social participation of children with atypical motor development?

Participants will answer two of three questionnaires:

* The Participation and Environment Measure - Children and Youth or the Young Children's Participation and Environment Measure, depending on the age of their child

.The Pediatric Evaluation of Disability Inventory - PEDI.

DETAILED DESCRIPTION:
The limitation in the execution of activities and tasks, as well as the restriction in the social participation of children considered atypical are considered biopsychosocial aspects of health according to the model of the International Classification of Disability and Health Functionality (ICF). The perception of the difficulties and limitations in the execution of the tasks, the barriers and facilitators of the environments and the participation and its restrictions, can be important to follow minimal or expressive improvements, indicate important changes in the environment and favor positive changes in the lives of children.

ELIGIBILITY:
Inclusion Criteria:

* Legal guardians of children aged up to 11 years and 11 months with motor disability
* Most be in Physio-therapeutic care at the School Clinic on the Realengo campus of the Federal Institute of Education, Science and Technology of Rio de Janeiro.

Exclusion Criteria:

* Guardians of children with a health condition associated with the Nervous System without motor limitations
* Other health conditions.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Legal guardians of children from 0 to 11 years and 11 months of age with clinical diagnosis of nervous system health conditions with motor limitations.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-10-07 (Actual); Primary Completion 2023-09-25 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Perception of caregivers/guardians of children with neuromotor disabilities regarding participation in three sections: home, school, and community. | 4 months
  Evaluated by PEM-CY and YC-PEM, each item on participation is evaluated in three dimensions: frequency (seven-point scale), involvement (five-point scale) and desire for change (scores from zero to 100%). The environment, in turn, is evaluated by its characteristics, as well as by the availability of services and resources (scores from zero to 100%).
Perception of caregivers/guardians of children with neuromotor disabilities regarding environmental factors that may be barriers or facilitators in three sections: home, school, and community. | 4 months
  Evaluated by PEM-CY and YC-PEM, each item on participation is evaluated in three dimensions: frequency (seven-point scale), involvement (five-point scale) and desire for change (scores from zero to 100%). The environment, in turn, is evaluated by its characteristics, as well as by the availability of services and resources (scores from zero to 100%).
Perception of caregivers/guardians of children with neuromotor disabilities about the child's performance in daily activities | 4 months
  Evaluated by PEDI, the score of Part I is the sum of the items scored with 1, that is, items that represent the ability to perform the activity. In Part II, each item can be scored between 0 and 5 points. Receives 5 the item in which the child performs the task independently and 0 when it needs full assistance. Scores 4 (supervision), 3 (minimum assistance), 2 (moderate assistance) and 1 (maximum assistance) represent the amount of help the child receives in the activities. These points are also added. Part 3 is qualitative.
Perception of caregivers/guardians of children with neuromotor disabilities about the child's mobility and the need for caregiver help | 4 months
  Evaluated by PEDI, the score of Part I is the sum of the items scored with 1, that is, items that represent the ability to perform the activity. In Part II, each item can be scored between 0 and 5 points. Receives 5 the item in which the child performs the task independently and 0 when it needs full assistance. Scores 4 (supervision), 3 (minimum assistance), 2 (moderate assistance) and 1 (maximum assistance) represent the amount of help the child receives in the activities. These points are also added. Part 3 is qualitative.
Perception of caregivers/guardians of children with neuromotor disabilities about the child's need for changes in the environment and in the child | 4 months
  Evaluated by PEDI, the score of Part I is the sum of the items scored with 1, that is, items that represent the ability to perform the activity. In Part II, each item can be scored between 0 and 5 points. Receives 5 the item in which the child performs the task independently and 0 when it needs full assistance. Scores 4 (supervision), 3 (minimum assistance), 2 (moderate assistance) and 1 (maximum assistance) represent the amount of help the child receives in the activities. These points are also added. Part 3 is qualitative.

CONTACTS AND LOCATIONS:
Overall Officials: Elisa B Van Eyken, PhD, Principal Investigator — Instituto Federal de Educação, Ciência e Tecnologia do Rio de Janeiro
Locations (1):
- Campus Realengo do IFRJ, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bosak DL, Jarvis JM, Khetani MA. Caregiver creation of participation-focused care plans using Participation and Environment Measure Plus (PEM+), an electronic health tool for family-centred care. Child Care Health Dev. 2019 Nov;45(6):791-798. doi: 10.1111/cch.12709. Epub 2019 Jul 30. PMID 31313843
- [Background] Burgess A, Boyd RN, Ziviani J, Ware RS, Sakzewski L. Self-care and manual ability in preschool children with cerebral palsy: a longitudinal study. Dev Med Child Neurol. 2019 May;61(5):570-578. doi: 10.1111/dmcn.14049. Epub 2018 Oct 7. PMID 30294776
- [Background] Coster W, Law M, Bedell G, Khetani M, Cousins M, Teplicky R. Development of the participation and environment measure for children and youth: conceptual basis. Disabil Rehabil. 2012;34(3):238-46. doi: 10.3109/09638288.2011.603017. PMID 21981404
- [Background] Krieger B, Schulze C, Boyd J, Amann R, Piskur B, Beurskens A, Teplicky R, Moser A. Cross-cultural adaptation of the Participation and Environment Measure for Children and Youth (PEM-CY) into German: a qualitative study in three countries. BMC Pediatr. 2020 Oct 24;20(1):492. doi: 10.1186/s12887-020-02343-y. PMID 33099320
- [Background] Thompson SV, Cech DJ, Cahill SM, Krzak JJ. Linking the Pediatric Evaluation of Disability Inventory-Computer Adaptive Test (PEDI-CAT) to the International Classification of Function. Pediatr Phys Ther. 2018 Apr;30(2):113-118. doi: 10.1097/PEP.0000000000000483. PMID 29498960
- [Background] Khetani MA, Albrecht EC, Jarvis JM, Pogorzelski D, Cheng E, Choong K. Determinants of change in home participation among critically ill children. Dev Med Child Neurol. 2018 Aug;60(8):793-800. doi: 10.1111/dmcn.13731. Epub 2018 Mar 25. PMID 29574916
- [Background] Mancini MC, Coster WJ, Amaral MF, Avelar BS, Freitas R, Sampaio RF. New version of the Pediatric Evaluation of Disability Inventory (PEDI-CAT): translation, cultural adaptation to Brazil and analyses of psychometric properties. Braz J Phys Ther. 2016 Nov-Dec;20(6):561-570. doi: 10.1590/bjpt-rbf.2014.0166. Epub 2016 Jun 16. PMID 27333475
- [Background] Miller AR, Rosenbaum P. Perspectives on "Disease" and "Disability" in Child Health: The Case of Childhood Neurodisability. Front Public Health. 2016 Oct 26;4:226. doi: 10.3389/fpubh.2016.00226. eCollection 2016. PMID 27833905
- [Background] Lexell J, Brogardh C. The use of ICF in the neurorehabilitation process. NeuroRehabilitation. 2015;36(1):5-9. doi: 10.3233/NRE-141184. PMID 25547759
- [Background] Bornbaum CC, Day AM, Izaryk K, Morrison SJ, Ravenek MJ, Sleeth LE, Skarakis-Doyle E. Exploring use of the ICF in health education. Disabil Rehabil. 2015;37(2):179-86. doi: 10.3109/09638288.2014.910558. Epub 2014 Apr 22. PMID 24754598
- See also: YC-PEM - Questionaire — http://canchild.ca/en/shop/23-yc-pem-young-children-s-participation-and-environment-measure

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-30): https://cdn.clinicaltrials.gov/large-docs/25/NCT06876025/Prot_SAP_000.pdf
  • Informed Consent Form (2023-07-30): https://cdn.clinicaltrials.gov/large-docs/25/NCT06876025/ICF_001.pdf